CLINICAL TRIAL: NCT01599832
Title: DCE-MRI as Pazopanib Biomarker in Metastatic Renal Cancer
Brief Title: Dynamic Contrast-Enhanced Magnetic Resonance Imaging in Measuring Effects of Pazopanib Hydrochloride in Patients With Metastatic Kidney Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-0121; NCI-2012-00676 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pazopanib hydrochloride, DCE-MRI) (Experimental): Patients receive pazopanib hydrochloride PO QD in the absence of disease progression or unacceptable toxicity. Patients undergo dynamic contrast-enhanced MRI at baseline, day 8, and prior to courses 3, 5, and 7.
  Interventions: Drug: pazopanib hydrochloride; Other: laboratory biomarker analysis; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Other: pharmacogenomic studies

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: laboratory biomarker analysis — Correlative studies
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Undergo dynamic contrast-enhanced magnetic resonance imaging
  Other Names: DCE-MRI
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study

SUMMARY:
The purpose of this study is to find out what effects pazopanib (pazopanib hydrochloride) (also called Votrient®) may have on MRI (magnetic resonance imaging) scans, blood pressure, and various proteins in the blood. Pazopanib is Food and Drug Administration (FDA) approved for treating renal cell cancer. It is an agent that prevents angiogenesis, which is new blood vessel formation. The use of pazopanib described in this study is a standard of care, but the additional MRI and blood tests that will be performed are experimental

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether a K^trans rise from nadir is predictive of subsequent tumor growth.

SECONDARY OBJECTIVES:

I. To determine the association between changes in mean ambulatory blood pressure measurements, K^trans, and tumor size changes with pazopanib therapy.

II. To determine the association between changes in soluble vascular endothelial growth factor receptor 2 (sVEGFR2) measurements, K^trans, and tumor size changes with pazopanib therapy.

TERTIARY OBJECTIVES:

I. To explore previously described single nucleotide polymorphisms (SNP's) as pharmacogenomic biomarkers.

II. To model tumor growth kinetics using radiologic tumor size measurements. III. To explore other serum and plasma based putative biomarkers of vascular endothelial growth factor (VEGF) pathway inhibition.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity. Patients undergo dynamic contrast-enhanced MRI at baseline, day 8, and prior to courses 3, 5, and 7.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up; procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* Histologically confirmed diagnosis of clear cell renal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Measurable disease at least 2 cm in the shortest dimension in the abdomen or pelvis
* No clinical contra-indication to contrast enhanced MRI
* No prior pazopanib therapy
* Archived tumor tissue must be provided for all subjects
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Hemoglobin >= 9 g/dL (5.6 mmol/L); subjects may not have had a transfusion within 7 days of screening assessment
* Platelets >= 100 X 10^9/L
* Total bilirubin =< 1.5 X upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 X ULN; concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN are not permitted
* Estimated glomerular filtration rate (GFR) (modification of renal disease [MDRD] equation) > 30 ml/min
* Urine protein to creatinine ratio (UPC) < 1; if UPC >= 1, then a 24-hour urine protein must be assessed; subjects must have a 24-hour urine protein value < 1 g to be eligible
* A female is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

  * A hysterectomy
  * A bilateral oophorectomy (ovariectomy)
  * A bilateral tubal ligation
  * Is post-menopausal

    * Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40 pg/mL (< 140 pmol/L)
    * Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
* Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception; acceptable contraceptive methods include:

  * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
  * Oral contraceptive, either combined or progestogen alone
  * Injectable progestogen
  * Implants of levonorgestrel
  * Estrogenic vaginal ring
  * Percutaneous contraceptive patches
  * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
  * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
  * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Not lactating; female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug

Exclusion Criteria:

* Prior malignancy; Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug; screening with CNS imaging studies (computed tomography [CT] or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment

Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

* Malabsorption syndrome
* Major resection of the stomach or small bowel

  * Presence of uncontrolled infection
  * Corrected QT interval (QTc) > 480 msecs using Bazett's formula
  * History of any one or more of the following cardiovascular conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Coronary artery bypass graft surgery
* Symptomatic peripheral vascular disease

  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
  * Poorly controlled hypertension (defined as systolic blood pressure (SBP) of >= 140 mmHg or diastolic blood pressure [DBP] of >= 90 mmHg); Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; blood pressure (BP) must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP/DBP values from each BP assessment must be < 140/90 mmHg in order for a subject to be eligible for the study
  * History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months; Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
  * Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
  * Evidence of active bleeding or bleeding diathesis
  * Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
  * Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug
  * Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
  * Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
  * Treatment with any of the following therapies:
* Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
* Anti-cancer chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment

  * Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity, except alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care (Peoria), Peoria, Illinois

REFERENCES:
- [Derived] Sweis RF, Medved M, Towey S, Karczmar GS, Oto A, Szmulewitz RZ, O'Donnell PH, Fishkin P, Karrison T, Stadler WM. Dynamic Contrast-Enhanced Magnetic Resonance Imaging as a Pharmacodynamic Biomarker for Pazopanib in Metastatic Renal Carcinoma. Clin Genitourin Cancer. 2017 Apr;15(2):207-212. doi: 10.1016/j.clgc.2016.08.011. Epub 2016 Aug 17. PMID 27634566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 63 [50 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
  African American | 2
  Hispanic | 2
  Not reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression
Description: Specifically, whether the change in K^trans (the rise from nadir) as a time-dependent covariate, as assessed by the method described in Donner, is associated with disease progression.Progression was assessed using Response Evaluation Criteria in Solid Tumors (Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum recorded since the treatment started OR the appearance of one or more new lesions OR unequivocal progression of existing non-target lesions)
Time Frame: 2 years
Population: The accrued sample size of n=20 did not permit further assessment (as described in the Outcome Measure Description) of the primary endpoint, so simply reporting the median progression-free survival here
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Number analyzed (Participants) | 20
weeks | 32.1 [7.6 to 79.6]

2. Secondary Outcome: Change in K^Trans From Baseline
Description: K^trans is a derived measure from dynamic contrast-enhanced magnetic resonance imaging that reflects perfusion rate and capillary permeability. The change is reported as the log-transformed ratio of K^trans value at follow-up/baseline.
Time Frame: Baseline and 1, 8, 16, and 24 weeks post-treatment
Population: Included those with a baseline K^Trans value and at least 1 K^trans value at follow-up
Measure: Mean (Standard Deviation); unit: unitless [log(ratio)]
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Number analyzed (Participants) | 17
unitless [log(ratio)]
  week 1 | -0.680 (0.729)
  week 8 | -1.049 (0.634)
  week 16 | -0.998 (0.757)
  week 24 | -0.755 (0.952)

3. Secondary Outcome: Changes in Blood Pressure From Baseline to Post-treatment
Time Frame: Baseline and 1 week post-treatment
Population: Data were not collected
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in sVEGFR2 From Baseline to Post-treatment
Time Frame: Baseline and 1 week post-treatment
Population: Data not collected
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Progression-free Survival
Description: Specifically, whether baseline K^trans is associated with progression-free survival. Progression was assessed using Response Evaluation Criteria in Solid Tumors (Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum recorded since the treatment started OR the appearance of one or more new lesions OR unequivocal progression of existing non-target lesions)
Time Frame: 2 years
Population: Included those with a baseline K^trans value
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Number analyzed (Participants) | 18
weeks | 32.1 [7.6 to 79.6]
Statistical Analysis 1: Comparison: Treatment (Pazopanib Hydrochloride, DCE-MRI); Test type: Other; p = 0.083, Regression, Cox — P-value was from test of significance of log-transformed baseline K^trans; Multivariate model with adjustment for prior treatment, and clinical prognostic index (good/intermediate/poor) (n=16 had complete data)

ADVERSE EVENTS:
Description: All serious adverse events are reported. For other adverse events, those that occurred in >5% of patients are reported.
Arm/Group | Treatment (Pazopanib Hydrochloride, DCE-MRI)
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pazopanib Hydrochloride, DCE-MRI) (N=20)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Muscle Weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Pain (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pazopanib Hydrochloride, DCE-MRI) (N=20)
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 11
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 5
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 13
Dysgeusia (Nervous system disorders) | 3
Fatigue (General disorders) | 13
Headache (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Proteinuria (Renal and urinary disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Hypercalcemia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 2
Weight loss (Investigations) | 2
Creatinine increased (Investigations) | 2
Platelet count decreased (Investigations) | 3
chronic kidney disease (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
White blood cell decreased (Investigations) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 3
Hair color change (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes